CLINICAL TRIAL: NCT02951754
Title: Methylphenidate in Adults With Attention Deficit/Hyperactivity Disorder
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100358
Record Dates: First submitted 2016-10-31; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Adults; treatment; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IR-MPH (Experimental): Immediate-release methylphenidate (IR-MPH) 10 mg two or three times daily with doses increasing weekly until symptom control
  Interventions: Drug: Immediate-release Methylphenidate

INTERVENTIONS:
Drug: Immediate-release Methylphenidate — Standard initial dose of 10 mg, twice or three times daily with doses increasing weekly until symptom control or occurrence of limiting adverse effects
  Other Names: Ritaline

SUMMARY:
Methylphenidate (MPH) is the first-line pharmacological treatment for adults with Attention-Deficit/Hyperactivity Disorder (ADHD). Nevertheless, there is considerable interindividual variability regarding the dose required, tolerability and response rates to MPH. The aim of this study is to address the clinical and genetic predictors of MPH treatment outcomes in ADHD.

DETAILED DESCRIPTION:
Methylphenidate (MPH) is the most prescribed psychostimulant for children and adults with Attention-Deficit/Hyperactivity Disorder (ADHD). Meta-analyses and systematic reviews have shown that MPH is safe and efficacious in attenuating the core symptoms of ADHD, promoting overall clinical improvement. However, many patients still do not show an appropriate clinical response to the MPH treatment and there is considerable interindividual variability regarding the dose required, tolerability and response rates to MPH. Therefore, it is essential to address the clinical and genetic predictors of MPH treatment outcomes in ADHD.

ELIGIBILITY:
Inclusion Criteria:

* White Brazilian of European descent
* Fulfillment of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, (DSM-IV) diagnostic criteria for ADHD
* Eligibility to immediate-release MPH (IR-MPH) treatment

Exclusion Criteria:

* Contraindication for IR-MPH use
* Current stimulant treatment
* Evidence of a clinically significant neurological disease that might affect cognition (e.g., delirium, dementia, epilepsy, head trauma, and multiple sclerosis)
* Current or past history of psychosis
* Estimated intelligence quotient score lower than 70

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2002-02; Primary Completion 2032-12 (Estimated); Study Completion 2032-12 (Estimated)

PRIMARY OUTCOMES:
Self-reported changes in severity of ADHD symptoms | 1yr
  Evaluated by Swanson, Nolan and Pelham Rating Scale - Version IV (SNAP-IV) adapted to adults.
  Assessment points at baseline, 6 weeks, 3 months, 6 months and 1 year of treatment

SECONDARY OUTCOMES:
Self-reported changes in severity of oppositional defiant disorder symptoms | 1yr
  Evaluated by Swanson, Nolan and Pelham Rating Scale - Version IV (SNAP-IV) adapted to adults.
  Assessment points at baseline, 6 weeks, 3 months, 6 months and 1 year of treatment
Psychiatrist's judgment of improvement of patient's symptoms | 1yr
  Evaluated by Clinical Global Impression - Improvement scale (CGI-I). Assessment points at baseline, 6 weeks, 3 months, 6 months and 1 year of treatment

OTHER OUTCOMES:
Maintenance of ADHD diagnosis | 1yr
  Assessed by Schedule for Affective Disorders and Schizophrenia for School-Age Children (K-SADS).
  Assessment points at baseline, 6 months and 1 year of treatment
Changes in side effects | 1yr
  Evaluated by Barkley's Stimulants Side Effects Rating Scale. Assessment points at baseline, 6 weeks, 3 months, 6 months and 1 year of treatment
Changes in measures of anxiety | 1yr
  Evaluated by Beck Anxiety Inventory (BAI). Assessment points at baseline, 6 months and 1 year of treatment
Changes in measures of depression | 1yr
  Evaluated by Beck Depression Inventory (BDI). Assessment points at baseline, 6 months and 1 year of treatment
Changes in scores of mood disorders | 1yr
  Evaluated by Mood Disorder Questionnaire (MDQ). Assessment points at baseline, 6 months and 1 year of treatment
Changes in insomnia problems | 1yr
  Evaluated by Insomnia Severity Index (ISI). Assessment points at baseline, 6 months and 1 year of treatment
Changes in scores of physical activity | 1yr
  Evaluated by International Physical Activity Questionnaires (IPAQ). Assessment points at baseline, 6 months and 1 year of treatment
Changes in measures of quality of life | 1yr
  Evaluated by Adult ADHD Quality of Life Questionnaire (AAQoL). Assessment points at baseline, 6 months and 1 year of treatment
Changes in measures of functional impairment in the main contexts of patient's life | 1yr
  Evaluated by Sheehan Disability Scale (SDS). Assessment points at baseline, 3 months, 6 months and 1 year of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eugênio H Grevet, MD, PhD, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Program on Attention-Deficit/Hyperactivity Disorder (PRODAH); Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Faraone SV, Spencer T, Aleardi M, Pagano C, Biederman J. Meta-analysis of the efficacy of methylphenidate for treating adult attention-deficit/hyperactivity disorder. J Clin Psychopharmacol. 2004 Feb;24(1):24-9. doi: 10.1097/01.jcp.0000108984.11879.95. PMID 14709943
- [Background] Epstein T, Patsopoulos NA, Weiser M. Immediate-release methylphenidate for attention deficit hyperactivity disorder (ADHD) in adults. Cochrane Database Syst Rev. 2014 Sep 18;(9):CD005041. doi: 10.1002/14651858.CD005041.pub2. PMID 25230710
- [Background] Castells X, Cunill R, Capella D. Treatment discontinuation with methylphenidate in adults with attention deficit hyperactivity disorder: a meta-analysis of randomized clinical trials. Eur J Clin Pharmacol. 2013 Mar;69(3):347-56. doi: 10.1007/s00228-012-1390-7. Epub 2012 Sep 16. PMID 22983311
- [Background] Retz W, Retz-Junginger P. Prediction of methylphenidate treatment outcome in adults with attention-deficit/hyperactivity disorder (ADHD). Eur Arch Psychiatry Clin Neurosci. 2014 Nov;264 Suppl 1:S35-43. doi: 10.1007/s00406-014-0542-4. Epub 2014 Sep 18. PMID 25231833
- [Background] Steele M, Jensen PS, Quinn DM. Remission versus response as the goal of therapy in ADHD: a new standard for the field? Clin Ther. 2006 Nov;28(11):1892-908. doi: 10.1016/j.clinthera.2006.11.006. PMID 17213010
- [Background] Swanson JM, Schuck S, Porter MM, Carlson C, Hartman CA, Sergeant JA, Clevenger W, Wasdell M, McCleary R, Lakes K, Wigal T. Categorical and Dimensional Definitions and Evaluations of Symptoms of ADHD: History of the SNAP and the SWAN Rating Scales. Int J Educ Psychol Assess. 2012 Apr;10(1):51-70. PMID 26504617
- [Background] Brod M, Johnston J, Able S, Swindle R. Validation of the adult attention-deficit/hyperactivity disorder quality-of-life Scale (AAQoL): a disease-specific quality-of-life measure. Qual Life Res. 2006 Feb;15(1):117-29. doi: 10.1007/s11136-005-8325-z. PMID 16411036
- [Background] Morin CM, Belleville G, Belanger L, Ivers H. The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep. 2011 May 1;34(5):601-8. doi: 10.1093/sleep/34.5.601. PMID 21532953
- [Background] Gomes-Oliveira MH, Gorenstein C, Lotufo Neto F, Andrade LH, Wang YP. Validation of the Brazilian Portuguese version of the Beck Depression Inventory-II in a community sample. Braz J Psychiatry. 2012 Dec;34(4):389-94. doi: 10.1016/j.rbp.2012.03.005. PMID 23429809
- [Background] Gorenstein C, Andrade L. Validation of a Portuguese version of the Beck Depression Inventory and the State-Trait Anxiety Inventory in Brazilian subjects. Braz J Med Biol Res. 1996 Apr;29(4):453-7. PMID 8736107